CLINICAL TRIAL: NCT05478642
Title: Influence of Psychological Status on the Results of Pain Treatment in Patients With Gunshot and Mine-explosive Wounds
Acronym: IPSRPTPGaM-EW
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Principal Investigator, Bogomolets National Medical University
Other Study IDs: 158 2022/23/05/
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain; Psychological Disorders
Keywords: Chronic pain, gunshot wounds, mine-explosive wounds, psychological disorders
MeSH Terms: conditions — Chronic Pain; Mental Disorders; Wounds, Gunshot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Interventions: Other: The Hospital Anxiety and Depression Scale.
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022
  Interventions: Other: The Hospital Anxiety and Depression Scale.

INTERVENTIONS:
Other: The Hospital Anxiety and Depression Scale. — The study was carried out on the basis of the National Military Medical Clinical Center "Main Military Clinical Hospital". All patients participated in Operation Joint Forces and received gunshot wounds during combat operations.
  A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv.
  Other Names: Mississippi PTSD scale (military version); Chaban Quality of Life Scale

SUMMARY:
82.1% of patients with gunshot and mine-explosive wounds and wounds during hostilities in Ukraine have negative results of pain treatment, which leads to its chronicity. Examining the effect of psychological status on pain management outcomes in these patients may improve their treatment outcomes.

DETAILED DESCRIPTION:
The influence of the amount of damage and operative interventions on the results of pain treatment in patients with gunshot and mine-explosive wounds at the stages of treatment needs to be studied, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions through the prism of psychological disorders have its features. Since in 82.1% of cases it is not possible to achieve a positive result of treatment, the data of our study will play an important role in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* availability gunshot and mine-explosive wounds

Exclusion Criteria:

* absence gunshot and mine-explosive wounds

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was carried out on the basis of the National Military Medical Clinical Center "Main Military Clinical Hospital". All patients participated in Operation Joint Forces and received gunshot wounds during combat operations.
  A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv.
Sampling Method: Non-Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  evaluation of the number of points
Didier Bouhassiraa DN4 | 12 months
  evaluation of the number of points
The Hospital Anxiety and Depression Scale | 12 months
  evaluation of the number of points
Chaban Quality of Life Scale | 12 months
  evaluation of the number of points
Mississippi PTSD scale (military version) | 12 months
  evaluation of the number of points

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share the results